CLINICAL TRIAL: NCT05877872
Title: Reduced-target Resection Compared With Full-target Resection After Induction Chemotherapy in Resectable Recurrent Nasopharyngeal Carcinoma: a Multicentre, Randomised, Open-label, Phase 3 Trial
Brief Title: Reduced-target Resection After Induction Chemotherapy in Resectable Recurrent Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); First People's Hospital of Foshan (Other); Zhongshan People's Hospital, Guangdong, China (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Deputy director, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2023-04-03
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Nasopharyngeal Carcinoma; De-escaltion Therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced-target resection group (Experimental): Patients receive surgery according to pSTV-post-IC and adjuvant immunotherapy.
  Interventions: Procedure: Reduced-target resection; Drug: Adjuvant immunotherapy
- Full-target resection group (Active Comparator): Patients receive surgery according to pSTV-pre-IC and adjuvant immunotherapy.
  Interventions: Procedure: Full-target resection; Drug: Adjuvant immunotherapy

INTERVENTIONS:
Procedure: Reduced-target resection — Patients receive surgery according to pSTV-post-IC.
  Arms: Reduced-target resection group
Procedure: Full-target resection — Patients receive surgery according to pSTV-pre-IC.
  Arms: Full-target resection group
Drug: Adjuvant immunotherapy — Toripalimab(240 mg d1) continually applied since 1-2 weeks after surgery until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, investigator decision, or 1 year.

SUMMARY:
The goal of this clinical trial is to compare efficacy of two different resection extension in patients with resectable recurrent nasopharyngeal carcinoma after induction chemotherapy. The main question it aims to answer is that whether tumor regress areas after induction chemotherapy required complete resection. Patients will be randomly assigned to receive reduced-target resection or full-target resection after induction chemotherapy. Researchers will compare these two groups to see if the efficacy of reduced-target resection is not inferior to full-target resection.

DETAILED DESCRIPTION:
Induction chemotherapy is often used preoperatively to reduce the size, extent, or stage of the tumor, thereby making the surgery more likely to be successful. However, there are still many patients with marginal recurrence after induction chemotherapy combined with surgery. With the progress of treatment methods, high efficient and low toxicity adjuvant immunotherapy is helpful to kill the minimal residual tumor lesions. Hence, whether complete resection is still necessary for areas with tumor regression after induction chemotherapy needs further investigation. Because of the organs at risk around the nasopharynx, any treatment strategy that can reduce the scope of tumor resection is of great significance. Therefore, by comparing reduced-target resection and full-target resection after induction chemotherapy, we aim to investigate whether reduced-target resection after induction chemotherapy is not inferior to full-target resection, but it greatly reduces the risk and difficulty of surgery. Even if marginal recurrence occurs after reduced-target resection, early intervention can still be performed through closely follow-up, without affecting the overall survival of patients.

When patients enroll this study, GTV-pre-IC (Gross Tumor Volume before induction chemotherapy) was defined according to the magentic resonance imaging before induction chemotherapy and GTV-post-IC (Gross Tumor Volume after induction chemotherapy) defined according to the magentic resonance imaging after induction chemotherapy. The pSTV-pre-IC (planing Surgical Tumor Volume before induction chemotherapy) and pSTV-post-IC (planing Surgical Tumor Volume after induction chemotherapy) were the GTV-pre-IC and GTV-post-IC plus an additional 0.5-1.0 cm peripheral mucosa margin and a 2-3 mm basal margin on the surface skull base. Patiens in experiment group will receive reduced-target resection, which resection extension is according to pSTV-post-IC. While patients in control group will receive full-target resection, which is according to pSTV-pre-IC. After surgery, the acturial resection area was defined as aSTV, which would be used for quality control. If aSTV does not cover pSTV, patients will be excluded in per-protocol set.

ELIGIBILITY:
Inclusion Criteria:

1. The recurrence time is more than 6 months from the end of radiotherapy.
2. Histologically confirmed recurrent nasopharyngeal carcinoma.
3. Resectable nasopharyngeal diseases: recurrent T1 (the tumor is confined in nasopharynx, oropharynx and/or nasal cavity without parapharyngeal involvement); recurrent T2 (the tumor is confined in the superficial parapharyngeal spacer and is more than 0.5cm far from the internal carotid artery) and recurrent T3 (the tumor is confined in the base wall of the sphenoid sinus and is more than 0.5cm far from the internal carotid artery and cavernous sinus) (according to the 8th edition of American Joint Committee on Cancer (AJCC) staging system for nasopharyngeal carcinoma). If the tumor invaded the internal carotid artery, or the instance from the internal carotid artery was less than 0.5cm, but the invasion area did not exceed the external edge of the internal carotid artery, the patients could be enrolled after internal carotid artery pretreatment (including internal carotid artery embolization or stent implantation).
4. After 3 cycles induction chemotherapy (Platinum based chemotherapy [gemcitabine/paclitaxel and platinum] and immunotherapy[PD-1/PD-L1 antibody] or a GAP regmen[gemcitabine, Apatinib and immunotherapy[PD-1/PD-L1 antibody]), patients achieved at least PR according to RECIST criteria, and the reduction of pSTV after induction chemotherapy more than 50%.
5. Given written informed consent.

Exclusion Criteria:

1. Karnofsky Performance Status (KPS) ≤70.
2. Has severe medical disorder, important organ dysfunction, and/or a substantial history of mental illness.
3. Tumor confined to the roof or the posterior wall of nasopharynx, without expected benefit from reduced-target resection.
4. Unresectable recurrent regional lymph node diseases (recurrent N1-3) with prevertebral fascia, cervical vertebrae, or common/internal carotid artery involvement (according to the 8th edition of AJCC staging system).
5. Clinically diagnosed with metastatic NPC.
6. Has known subjects with other malignant tumors (except for cured skin basal cell carcinoma or cervical carcinoma in situ).
7. Received a systematic or local glucocorticoid therapy within 4 weeks of planned start of study treatment.
8. Suffered from diseases need long-term treatment with immunosuppressive drugs, or required systematic or local glucocorticoid therapy with immunosuppressive doses.

   Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) agent.
9. Has active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy). Patients with skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) will be allowed to enroll.
10. Has a known history of human immunodeficiency virus (HIV), has hepatitis B surface antigen (HBsAg) positive with hepatitis B virus (HBV) DNA copy number of ≥1000cps/ml or hepatitis C virus (HCV) antibody positive.
11. Has received a live vaccine within 4 weeks of planned start of study treatment. Pregnancy or breast feeding.
12. Cannot complete regular follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 3 years
  Overall survival is calculated from the date of randomization to the date of death of any cause, censored on the last date of known survival if no death has happened

SECONDARY OUTCOMES:
The incidence of Severe Adverse events | 3 years
  The incidence of severe adverse events was defined as the incidence of grade 3 or worse adverse event, including acute and late toxicities.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) overall | 3 years
  The quality of life was assessed per EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0).
In-field recurrence rate | 3 years
  The rate of recuurence within the Gross Tumor Volume before induction chemotherapy
Progression-free survival (PFS) | 3 years
  Progression-free survival is calculated from the date of randomization to the date of death of any cause or the first progress at any site, censored on the last date of tumor evaluation if no progress has happened.
Loco-regional relapse-free survival (LRRFS) | 3 years
  The event for loco-regional relapse-free survival (LRRFS) was loco-regional recurrence. The duration was calculated from the date of treatment initiation to the date of loco-regional relapse or last follow-up.
Distant metastasis-free survival (DMFS) | 3 years
  The event for distant metastasis-free survival (DMFS) was distant metastasis. The duration was calculated from the date of treatment initiation to the date of distant metastasis or the last follow-up.
The proportion of Internal carotid artery pretreatment | 1 Day of surgery
  the proportion of the patients who received Internal carotid artery pretreatment (including endoscopic-assisted transcervical protection of the parapharyngeal ICA, embolization, stent implantation and so on).
Surgery-related adverse event | 3 years
  The incidence of surgey-related adverse events, including operative accidents and complications.
Operative resection time | 1 Day of surgery
  Time from making mucosa incision to completely resecting the tumor.
Estimated blood loss | 1 Day of surgery
  Blood loss will be measured according to the suction and the weight of wet gauze, and then minus the irrigation.
Progression-free survival after salvage treatment as assessed by the investigator (PFS2) | 3 years
  The time from randomization to second/subsequent disease progression after initiation of new anticancer therapy, or death from any cause, which occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China